CLINICAL TRIAL: NCT00614250
Title: A Double-blind, Randomized, Placebo-controlled, Study of the Safety and Activity of Four Escalating Single Doses of AVE0657 in Patients Suffering From Obstructive Sleep Apnea Hypopnea Syndrome
Brief Title: Evaluation of the Effect of AVE0657 on Obstructive Sleep Apnea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT6796; EudraCT 2007-002174-58
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2009-07-20 (Estimated); Status verified 2009-07

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Dose Level 1 (Experimental)
  Interventions: Drug: AVE0657
- Dose Level 2 (Experimental)
  Interventions: Drug: AVE0657
- Dose Level 3 (Experimental)
  Interventions: Drug: AVE0657
- Dose Level 4 (Experimental)
  Interventions: Drug: AVE0657
- Placebo (Placebo Comparator): 12 subjects: 3 subjects per dose level
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: AVE0657 — capsules once a day at bedtime
  Arms: Dose Level 1; Dose Level 2; Dose Level 3; Dose Level 4
Drug: placebo — capsules once a day at bedtime
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the activity of 4 escalating doses of AVE0657 in comparison to placebo in patients with Obstructive Sleep Apnea Hypopnea Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with Obstructive Sleep Apnea Hypopnea Syndrome based on International Classification of Sleep Disorders

Exclusion Criteria:

* Subjects having been treated by Continuous Positive Airway Pressure, oral appliance during 4-weeks prior to randomization
* Chronic respiratory disease or inadequate respiratory parameters
* Body Mass Index (BMI) of ≤20 kg/m² or ≥35 kg/m²
* Surgical procedure to correct apnea within the last three months.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Change in Apnea Hypopnea Index (AHI) | 2 days

SECONDARY OUTCOMES:
Safety and tolerability | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Patrick LEVY, Professor, Principal Investigator — Hôpital Michallon - Grenoble - France
Locations (3):
- Sanofi- Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Barcelona, Spain